CLINICAL TRIAL: NCT03073642
Title: Effects of Pain Therapeutic Education and Hydrotherapy on Pain, Depression, Anxiety, Quality of Life and Quality of Sleep of Women With Fibromyalgia
Brief Title: Effects of Pain Therapeutic Education and Hydrotherapy on Physical Function, Pain and Sleep of Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Mariana Arias Avila, Principal Investigator, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFSCarFMS; 2017/03278-0 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2017-02-20; First posted 2017-03-08 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Fibromyalgia
Keywords: Hydrotherapy; Pain education
MeSH Terms: conditions — Fibromyalgia | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial with 1:1 allocation
Who Masked: Care Provider, Investigator
Masking Description: Outcomes assessor will not know in which group volunteers are allocated; Care provider will not know outcome measures for any volunteers before study completion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrotherapy (Active Comparator): Patients allocated to this group will perform 12 weeks of hydrotherapy treatment, with global exercises. Hydrotherapy sessions will last 45 minutes and will be performed twice a week.
  Exercises will involve aerobic exercises (in the pool) with exercises for upper and lower limbs, and trunk.
  Interventions: Other: Hydrotherapy
- Hydrotherapy and Pain Education (Experimental): Patients allocated to this group will perform 12 weeks of hydrotherapy treatment, with global exercises. Hydrotherapy sessions will last 45 minutes and will be performed twice a week.
  Exercises will involve aerobic exercises (in the pool) with exercises for upper and lower limbs, and trunk.
  During the 12 weeks of hydrotherapy treatment, volunteers will also receive 4 sessions of Pain Therapeutic Education, which is also known as Pain Neuroscience Education, which involves patient education on pain neurophysiology, pain chronification and amplification mechanisms, and chronic pain management. These sessions will be performed in specific dates scheduled according to the volunteers' availability, and with intervals that can last from one to two weeks.
  Interventions: Other: Pain Education; Other: Hydrotherapy

INTERVENTIONS:
Other: Pain Education — Together with hydrotherapy, patients will receive pain therapeutic education
  Other Names: Pain Neuroscience Education, Pain Therapeutic Education
  Arms: Hydrotherapy and Pain Education
Other: Hydrotherapy — Hydrotherapy sessions, lasting 45 minutes, twice a week for 12 weeks.

SUMMARY:
Fibromyalgia (FM) is a prevalent and disabling disease, that affects mostly women and its main characteristic is chronic pain. Several studies have shown that hydrotherapy is effective in the improvement of symptoms and quality of life of this population; other studies have shown that Pain Therapeutic Education (PTE) is also effective in this sense. PTE is one cheap, easy to apply intervention, with very positive results in chronic pain situations. However, there is a lack of studies that have shown the effects of this intervention on FM. Hence, this study will aim to verify the effectiveness of the hydrotherapy and PTE on women with FM. Sixty women will be randomly allocated in two groups: hydrotherapy and hydrotherapy + PTE. Before treatment start, the investigators will evaluate pain (visual analogue scale, presence of myofascial trigger points and pressure pain threshold over the scalene, upper trapezius, infraspinatus, piriformis, iliopsoas and soleus, bilaterally), quality of life (Fibromyalgia Impact Questionnaire and medical outcomes study 36-item short-form health survey), depression (Beck Depression Inventory), anxiety (Beck Anxiety Inventory) and sleep quality (Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale). Hydrotherapy treatment will last 12 weeks. Women will be evaluated other 3 times: after 6 and 12 weeks (treatment middle and end) and 12 weeks after treatment completion (follow-up). Women in the hydrotherapy group will receive a folder with explanations on FM. Women in the hydrotherapy + PTE will participate of 4 meetings over 12 treatment weeks, in which themes like pain physiology, pain chronification and exacerbation and pain self-management, as well as information on FM will be approached. Statistical analysis will include qualitative and quantitative variable description. Correlation among variables will also be analyzed. Level of significance will be set at 5%.

DETAILED DESCRIPTION:
The investigators will select at least 80 women with fibromyalgia (FM) for this study, in which pain (through pressure pain threshold and number of active myofascial trigger points), quality of life, FM impact on quality of life and function, depression, anxiety and quality of sleep will be evaluated.

After evaluating the volunteer, the participant will be randomly allocated to one of two groups: hydrotherapy treatment (HT), and hydrotherapy treatment together with pain therapeutic education (HT+PTE).

All volunteers will perform 12 weeks of hydrotherapy treatment, in which the investigators will perform global exercises for upper and lower limbs and trunk.

Volunteers in the HT+PTE group will receive, throughout the 12 weeks of HT, 4 sessions of PTE, in which the investigators will teach pain neurophysiology, pain chronification and pain management.

Evaluation sessions will take place before treatment, after 6 and 12 weeks of HT and after 12 weeks of treatment ending.

In all evaluations sessions, the investigators will collect data on those aspects previously described.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and medical Fibromyalgia Diagnosis according to ACR Diagnostic criteria 2010 and 2016;
* Willing to perform hydrotherapy as treatment.

Exclusion Criteria:

* Cognitive deficits that prevent volunteers from understanding evaluation and treatment procedures;
* Uncontrolled systemic illnesses (diabetes, hypertension);
* Neurological and musculoskeletal conditions that may interfere in the evaluation and treatment procedures (palsies, sensitivity alterations, advanced osteoarthritis);
* Infecto-contagious illnesses (especially in the urinary tract);
* Alcohol or drug abuse;
* Pregnancy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Changes in Pain throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Visual Analogue Scale (VAS - 100mm) for pain

SECONDARY OUTCOMES:
Changes in number of active myofascial trigger points throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Number of active myofascial trigger points
Changes in depression throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Depression clinical symptoms (measured through Hospital Anxiety and Depression Scale)
Changes in anxiety throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Anxiety clinical symptoms (measured through Hospital Anxiety and Depression Scale)
Changes in Impact of Fibromyalgia in Quality of life throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Quality of life measured through Revised Fibromyalgia Impact Questionnaire
Changes in Quality of life throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Quality of life measured through questionnaire Medical Outcomes Sudy 36-item Short-Form Health Survey (sf-36)
Changes in Sleep throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Sleep quality measured through two questionnaires: Pittsburgh Quality of Sleep Index and Epworth Sleepiness Scale
Changes in Pain neurophysiology learning throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  For the Pain Therapeutic Education group, index of Pain Neurophysiology learning with an specific questionnaire
Changes in knowledge of Fibromyalgia throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Fibromyalgia Knowledge will be measured through Fibromyalgia Knowledge Questionnaire
Changes in Appraisal of Self-Care Agency throughout time | Before treatment, after 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Appraissal of Self-Care Agency through The Appraisal of Self-Care Agency Scale - Revised (ASAS-R) scores
Pacient satisfaction with the intervention | After 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Structured questionnaire through which patient will answer about satisfaction with treatment, with a 5-point Likert Scale, with the possible asnswers: "Totally Agree", "Agree", "Neutral", "Disagree" and "Totally Disagree", relative to the following affirmations: 1) I am satisfied with the treatment I received; 2) I believe this treatment was helpful for my condition; 3) I believe my health status has improved after treatment; 4) I will include in my daily life activities things I have learned during my treatment; 5) I will recommend this treatment to someone who has the same health condition as me.
Patient's perception of change | After 6 and 12 weeks of treatment and after 12 weeks of treatment completion.
  Self-perception of change with the Global Rating of Change Scale; with this scale from -7 to 7, the participant will rate her perception of change after intervention. The negative values will be considered as a worsening in the health status, and the positive values, as a improvement in the health condition of the participant. Zero will be considered as no change in the health status.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana A Avila, Ph.D., Principal Investigator — UFSCar
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
All results shall be disclosed in a form that no individual volunteers shall be identified.

REFERENCES:
- [Background] Queiroz LP. Worldwide epidemiology of fibromyalgia. Curr Pain Headache Rep. 2013 Aug;17(8):356. doi: 10.1007/s11916-013-0356-5. PMID 23801009
- [Background] Ortega E, Bote ME, Giraldo E, Garcia JJ. Aquatic exercise improves the monocyte pro- and anti-inflammatory cytokine production balance in fibromyalgia patients. Scand J Med Sci Sports. 2012 Feb;22(1):104-12. doi: 10.1111/j.1600-0838.2010.01132.x. Epub 2010 Jun 1. PMID 20536907
- [Derived] Sousa AP, Almeida LA, Lourenco BP, Alvares LD, Avila MA. Pain neuroscience education improves quality of life when added to aquatic exercise therapy for women with fibromyalgia: randomized controlled clinical trial. Disabil Rehabil. 2024 Apr;46(8):1559-1569. doi: 10.1080/09638288.2023.2201510. Epub 2023 Apr 18. PMID 37070715